CLINICAL TRIAL: NCT04789278
Title: Incidental Coronary Calcification Quality Improvement Project
Acronym: ICC QI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexander Sandhu, Principal Investigator, Instructor of Medicine, Division of Cardiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICC-QI-2021
Record Dates: First submitted 2021-02-26; First posted 2021-03-09 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Atherosclerotic Cardiovascular Disease; Coronary Artery Disease
Keywords: Coronary Calcium; Statin; Non-gated Chest CT
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Notification (Experimental): Patients randomized to notification will receive a message sent by either the electronic health record (EHR) patient portal or postal mail that will inform them of the CAC identified on their previous chest CT. It will provide an overview of CAC, an image of their chest CT, and a recommendation that they discuss this finding with their clinician. These clinicians will be notified of these findings via an earlier EHR message. Any treatment decisions will be made by the patient and their clinician.
  Patients randomized to notification who are not prescribed a statin medication and do not have a documented discussion regarding statin therapy within three months will be sent a second message at that time. Their primary care providers will receive a second EHR message concurrently.
  Interventions: Other: Notification
- Usual Care (No Intervention): Both arms have previously had their CT scans reported according to standard clinical practice. This may include notification of the CAC in the imaging report. The usual care arm will not receive any additional notification beyond this standard of care during the project.

INTERVENTIONS:
Other: Notification — Notification of coronary calcium to the patient and their clinician
  Arms: Notification

SUMMARY:
This is a multi-center, randomized quality improvement project. At least 200 statin-naïve patients without a history of atherosclerotic cardiovascular disease with incidental coronary artery calcium (CAC) on a prior non-gated chest CT will be enrolled across the Stanford Healthcare System and the Palo Alto Veteran's Affairs Healthcare System. Patients will be randomized in a 1:1 fashion to notification or usual care arms. The primary aim of this project is to estimate the increase in 6-month statin prescription among statin-naïve patients without a history of atherosclerotic cardiovascular disease with incidental CAC on a non-gated chest CT who are randomized to receive notification of their findings vs. usual care.

ELIGIBILITY:
Inclusion Criteria:

* Non-gated chest CT between 2014-2019
* The presence of CAC confirmed by manual review by an experienced radiologist
* Stanford affiliated primary care provider or endocrinologist for Stanford healthcare system patients and VA primary care provider for VA patients with at least 1 encounter since 2018

Exclusion Criteria:

* Current or prior statin or PCSK9 inhibitor therapy
* Prior diagnosis of ASCVD (coronary artery disease, peripheral arterial disease, cerebrovascular disease, coronary/peripheral revascularization)
* Prior coronary imaging (cardiac CT, invasive coronary angiography)
* Dementia
* Metastatic cancer or active cancer undergoing chemotherapy
* History of medical nonadherence

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Rate of Statin Prescription | Within 6 months
  Proportion of patients prescribed a statin

SECONDARY OUTCOMES:
Statin Intensity | 6 months
  Proportion of patients prescribed a high intensity, intermediate intensity, and low intensity statin
Total Cholesterol Level | 6 months
LDL Cholesterol Level | 6 months
HDL Cholesterol Level | 6 months
Triglyceride Level | 6 months
Systolic Blood Pressure | 6 months
Number of Hypertension Medications | 6 months
Hemoglobin A1c Level | 6 months
Body Mass Index | 6 months
Pooled cohort equations estimated 10-year risk of atherosclerotic cardiovascular disease | 6 months
Rate of Aspirin Prescription | 6 months
  Proportion of patients prescribed aspirin
Number of primary Care Clinical Encounters | 6 months
Number of Cardiology Referrals | 6 months
Number of Cardiovascular Diagnostic Tests | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T Sandhu, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital & Clinics, Stanford, California, United States

REFERENCES:
- [Derived] Sandhu AT, Rodriguez F, Ngo S, Patel BN, Mastrodicasa D, Eng D, Khandwala N, Balla S, Sousa D, Maron DJ. Incidental Coronary Artery Calcium: Opportunistic Screening of Previous Nongated Chest Computed Tomography Scans to Improve Statin Rates (NOTIFY-1 Project). Circulation. 2023 Feb 28;147(9):703-714. doi: 10.1161/CIRCULATIONAHA.122.062746. Epub 2022 Nov 7. PMID 36342823

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT04789278/Prot_SAP_000.pdf